CLINICAL TRIAL: NCT04340752
Title: Optimal Dosing of IC-Green for Visualization of Rotator Cuff Vascularity Using Advanced Imaging Modality Arthroscopy: A Prospective, Randomized Trial
Brief Title: Optimal Dosing of IC-Green for Visualization of Rotator Cuff Vascularity Using Advanced Imaging Modality Arthroscopy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-01995
Record Dates: First submitted 2020-04-02; First posted 2020-04-09 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Indocyanine Green

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1:ICG 7.5 mg (Experimental): Subjects in this group are randomized to receive 7.5 mg dose of Indocyanine Green (ICG) intravenously during the clinical surgery. ICG is a substance that binds to proteins in the blood and allows surgery teams to view blood vessels with greater precision.
  Interventions: Drug: Indocyanine Green
- Group 2:ICG 12.5 mg (Experimental): Subjects in this group are randomized to receive 12.5 mg dose of Indocyanine Green (ICG) intravenously during the clinical surgery. ICG is a substance that binds to proteins in the blood and allows surgery teams to view blood vessels with greater precision.
  Interventions: Drug: Indocyanine Green
- Group 3: ICG 25 mg (Experimental): Subjects in this group are randomized to receive 25 mg dose of Indocyanine Green (ICG) intravenously during the clinical surgery. ICG is a substance that binds to proteins in the blood and allows surgery teams to view blood vessels with greater precision.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — ICG is an injectable fluorescent pigment that binds to proteins in the blood and allows surgery teams to view blood vessels with greater precision. The ICG will not affect the course of the operative or postoperative period, and will be injected intravenously prior to the actual repair

SUMMARY:
Rotator cuff re-tear is a common delayed complication of arthroscopic rotator cuff repair. This process of re-tear is multifactorial and there has not been any readily identifiable perioperative measure that is predictive of subsequent rotator cuff failure. There have been no human studies looking at intraoperative assessment of rotator cuff vascularity, nor the predictive value that vascularity may have for rotator cuff re-tear. Indocyanine Green (ICG) has been safely used in patients for visualization purposes and has real potential for identifying vascularity in arthroscopic surgical patients. The aim of this study is to establish a standard dosing protocol for ICG in the arthroscopic visualization of rotator cuff vascularity.

DETAILED DESCRIPTION:
The primary study objective is to determine optimal dosing of an intravenous fluorescence solution (IC-Green) for arthroscopic evaluation of rotator cuff vascularity. The primary endpoint is surgeon's ability to assess vascularity within the rotator cuff based on a 5-point likert scale. The likert values from each of the three doses will undergo an ANOVA test to compare means of the three doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients has full or partial thickness rotator cuff tear and is scheduled to undergo arthroscopic rotator cuff repair
* Patient is at least 18 years of age and less than 80 years of age

Exclusion Criteria:

* Patient is less than 18 years of age or greater than 79 years of age
* Patient has a documented allergy to iodides
* Patients who have had iodide based radiology studies within the last seven (7) days prior to surgery
* Patient is pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Optimal dosing of an intravenous fluorescence solution (ICG) for arthroscopic evaluation of rotator cuff vascularity | up to 6 months post operative visit
  Advanced Imaging Modality (AIM) arthroscopy videos for each dosing arm will be collected and five signal intensity readings will be collected from the rotator cuff within each video. The ability to visualize rotator cuff vascularity will be graded by surgeons blinded to the ICG dosing using a 5 point Likert scale where 1 indicates worst visibility and 5 indicates best visibility. Post-hoc ANOVA analysis of surgeons' responses to determine what dose of ICG is optimal for the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Campbell, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to kirk.campbell@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.